CLINICAL TRIAL: NCT05676892
Title: Effects of Intravenous Ibuprofen on Acute Pain After Laparoscopic Cholecystectomy; a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Effects of Intravenous Ibuprofen on Acute Pain After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seoul_S11
Record Dates: First submitted 2022-12-28; First posted 2023-01-09 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Cholecystitis/Cholelithiasis
Keywords: ibuprofen; postoperative pain
MeSH Terms: conditions — Cholecystitis; Cholelithiasis; Pain, Postoperative | interventions — Cholecystectomy, Laparoscopic; Hematologic Tests; Blood Chemical Analysis; Urination; Blood Coagulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The experimental group in benign gallbladder disease (Experimental): inclusion criteria
  * Patients who underwent elective gallbladder surgery (cholelithiasis, chronic cholecystitis, gallbladder polyps, gallbladder adenomyomatosis) ② Patients between the ages of 19 and 65 ③ A person who voluntarily signed a written consent form after hearing and understanding the explanation of this clinical trial
  intravenous ibuprofen 800mg/8ml was used after surgery.
  Interventions: Procedure: Laparoscopic cholecystectomy
- The controled group in benign gallbladder disease (Experimental): inclusion criteria
  * Patients who underwent elective gallbladder surgery (cholelithiasis, chronic cholecystitis, gallbladder polyps, gallbladder adenomyomatosis) ② Patients between the ages of 19 and 65 ③ A person who voluntarily signed a written consent form after hearing and understanding the explanation of this clinical trial
  normal saline (Isotonic Sodium Chloride Injection Daihan(50mL/bag)) was used after surgery.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Method of operation
  1. Surgery was started under general anesthesia
  2. A trocar of 10 mm was placed on the navel, 5 mm under the blade, and a 5 mm trocar was placed on the right upper abdomen.
  3. Pneumoperitoneum was performed using CO2 gas in the abdominal cavity.
  4. Dissection started from Calot's triangle, and the operation was performed by retrograde cholecystectomy.
  5. The excised gallbladder was placed in a laparoscopic pocket and extracted through the umbilicus.
  6. The trocar was removed, and the skin was sutured
  Other Names: hematology, blood chemistry, urine, blood clotting, and chest x-rays were performed

SUMMARY:
This clinical trial is a medical intervention study to evaluate the necessity and effectiveness of intravenous ibupropan for postoperative acute pain relief after laparoscopic cholecystectomy in benign gallbladder disease. Comparison and evaluation of changes in pain scores after surgery according to the presence or absence of use.

DETAILED DESCRIPTION:
Cholecystectomy is the most common abdominal surgical procedure and is usually performed laparoscopically. Laparoscopic cholecystectomy is considered the standard surgery for gallstone disease, and this procedure has the advantages of less postoperative pain, better cosmetic results, shorter hospital stay, and faster wound healing than open cholecystectomy.

There are several factors that can cause pain after laparoscopic cholecystectomy, including stimulation of the phrenic nerve due to CO2 injection into the abdominal cavity, incision pain at the port site, and pain at the gallbladder removal site. Postoperative pain is an acute sensation that accompanies the surgical trauma and the observed inflammatory process and decreases as the tissue heals.

Postoperative analgesics are known to prevent pain-related effects in patients after surgery, such as increased cardiovascular system workload and increased stress response due to neuroendocrine and sympathetic nervous system activation. Like other NSAIDs, ibupropan is a propionic acid derivative that has anti-inflammatory, antipyretic and analgesic effects. The oral form has been used safely for a long time and is one of the most commonly used NSAIDs. Ibuprofan in the intravenous (IV) form has been used in the United States since 2009 for the treatment of mild to moderate and severe pain in combination with narcotic analgesics. Research on ibuprolan for intravenous injection is still insufficient, and there are very few studies showing its effect on pain relief after surgery. Therefore, this study was conducted in a double-blind, prospective, randomized, placebo-controlled clinical trial to investigate the evidence for clinical usefulness of the effect of intravenous ibupropan on postoperative pain in patients who underwent laparoscopic cholecystectomy.

Study population

1. Inclusion criteria

   ① Patients who underwent elective gallbladder surgery (cholelithiasis, chronic cholecystitis, gallbladder polyps, gallbladder adenomyomatosis)

   ② Patients between the ages of 19 and 65

   ③ A person who voluntarily signed a written consent form after hearing and understanding the explanation of this clinical trial
2. Exclusion criteria

   * Patients with acute cholecystitis

     ② Gallbladder cancer
   * Cholecystitis with a gallbladder thickness of 4 mm or more on CT or ultrasound

     * Cholecystitis with adhesions with surrounding organs due to inflammation of the gallbladder

       * Pregnant or lactating women

         ④ Those who undergo surgery at the same time due to other organ diseases

         ⑤ Those with immunosuppression and hemorrhagic tendencies

         ⑥ Persons who have undergone preoperative percutaneous cholecystectomy (PTGBD)

         ⑦ Persons who need drainage tube installation during surgery

         ⑧ Those who participated in other clinical trials within 3 months before screening

         ⑨ Persons judged by other investigators to be inappropriate to participate in this clinical trial
3. Target number of subjects and calculation basis In order to calculate the number of subjects in this study, it was assumed that the baseline postoperative pain score was the same in both groups based on the existing literature, and the VAS score within 6 hours after surgery was 2.33 ± 0.99 in the ibuprofen group and 3.20 ± 1.83 in the placebo group. seemed As a result of calculating the study subjects with 95% power using two-group T-test with two-side with a two-sided significance level of 0.05, each group requires 63 subjects, and calculating a 10% dropout rate, 70 subjects per group, a total of 140 subjects subject is required

Study design

1. Design of clinical trials This clinical trial is an exploratory clinical trial to evaluate whether intravenous analgesic use after surgery can help reduce postoperative pain scores in gallbladder disease requiring elective surgery. implement On the day of surgery, after determining whether the selection/exclusion criteria are met, suitable subjects are randomly assigned to the test group and control group in a 1:1 ratio. Only for the test group, an investigational drug (ibuprofen 800mg/8ml) is administered through intravenous injection after surgery, and physiological saline is administered for 30 minutes to the control group. Painkillers and physiological saline are administered repeatedly at 12-hour intervals from the first dose until the patient is discharged.

   On the day of surgery (OP day) and the day of discharge, an adverse reaction investigation, laboratory test, and physical examination are conducted to evaluate safety and efficacy, and the degree of postoperative pain and hospitalization period are evaluated. At 1 week after discharge, an outpatient visit is conducted for adverse events, laboratory tests, and physical examinations to evaluate the degree of postoperative pain, postoperative infection-related complications, complications other than infection, and whether additional procedures are required. In addition, when visiting the emergency room due to postoperative infection-related complications within one month after discharge, the degree of postoperative pain, rehospitalization, complications other than infection, and whether additional procedures are required are evaluated and compared.
2. Method of subject registration and randomization Subjects who have listened to the explanation of this clinical trial and agreed to voluntarily participate in the trial will be given a subject identification code in the order in which they signed the consent form at the screening visit. Randomization is performed to ensure the scientific validity of clinical trials by ensuring that the subjectivity of the investigator is not involved in the assignment.

Block randomization is performed to divide the patients into 2 groups and allocate them in a 1:1 ratio for patients who satisfy the selection/exclusion criteria and agree to participate in the clinical trial. For randomization, a statistician independent of this clinical trial generates a randomization number using SAS ver.9.4 for Microsoft Windows (SAS Institute Inc, NC, Cary, USA) or higher and assigns them sequentially.

Method of operation

1. Surgery was started under general anesthesia
2. A trocar of 10 mm was placed on the navel, 5 mm under the blade, and 5 mm trocar was placed on the right upper abdomen.
3. Pneumoperitoneum was performed using CO2 gas in the abdominal cavity.

   * Double pressure through CO2 gas was maintained at 12mmHg / and 2L / min.
4. Dissection started from Calot's triangle, and the operation was performed by retrograde cholecystectomy.

   * The cystic duct was ligated with a 10mm clip, and the cystic artery was also ligated with a 10mm clip.
   * If the cystic duct was unstably ligated, ligation was performed through an end loop.
   * After ligation, the gallbladder was dissected from the liver.
5. Washed the surgical site.
6. The excised gallbladder was placed in a laparoscopic pocket and extracted through the umbilicus.
7. The trocar was removed, the skin was sutured, and the operation was completed.

characteristics of observational and clinical test

* Hematology tests: Hematocrit, Hemoglobin, Platelet, WBC & Differential count
* Blood coagulation test: PT INR, aPTT, BT
* Blood chemistry test: SGOT (AST), SGPT (ALT), alkaline phosphatase, γ-GTP, bilirubin (total / direct), fasting plasma glucose, BUN, creatinine, sodium, potassium, chloride, total protein, albumin, uric acid, CPK, LDH, CRP
* Imaging medical examination
* Postoperative hospital stay
* Check for infection.
* Check for leakage of bile.
* Surgery time and bleeding amount were described.
* Postoperative complications

Statistical analysis In the case of categorical variables for the length of stay, surgical time, and complication data obtained as secondary endpoints, n (%) was presented, and the ratio difference between the two groups was tested using Chi-square or Fisher's exact test. In addition, for continuous variables, the mean, standard deviation, median, minimum, and maximum values were presented. The normality test was performed to test with Student's t-test for normal distribution and the non-normal distribution Wilcoxon rank-sum test. The difference between the two groups would be tested. All statistical analyses would use SPSS version 21.0, and it would be judged that it was statistically significant below the significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective gallbladder surgery (cholelithiasis, chronic cholecystitis, gallbladder polyps, gallbladder adenomyomatosis)

  * Patients between the ages of 19 and 65 ③ A person who voluntarily signed a written consent form after hearing and understanding the explanation of this clinical trial

Exclusion Criteria:

* Patients with acute cholecystitis

  ② Gallbladder cancer
* Cholecystitis with a gallbladder thickness of 4 mm or more on CT or ultrasound

  * Cholecystitis with adhesions with surrounding organs due to inflammation of the gallbladder

    * Pregnant or lactating women

      * Those who undergo surgery at the same time due to other organ diseases ⑤ Those with immunosuppression and hemorrhagic tendencies

        * Persons who have undergone preoperative percutaneous cholecystectomy (PTGBD)

          * Persons who need drainage tube installation during surgery ⑧ Those who participated in other clinical trials within 3 months before screening ⑨ Persons judged by other investigators to be inappropriate to participate in this clinical trial

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS (Visual Analogue Scale) score | 7 days
  Postoperative pain score in patients who underwent a laparoscopic cholecystectomy with the ibuprofen and normal saline.
  pain score : minimum 0 to maximum 10 (0:no pain - 10: worst pain)

SECONDARY OUTCOMES:
consumption of analgesics | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  consumption of analgesics after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sung eun Park, Study Director — The Catholic University of Korea
Locations (1):
- Department of HBP Surgery, Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

IPD SHARING:
Plan to Share IPD: No